CLINICAL TRIAL: NCT04226794
Title: Effect of Nutritional Counseling Associated With Transcranial Direct-current Stimulation in Binge Eating Reduction: A Single-blinded, Randomized Clinical Trial in Parallel With Simulated Use
Brief Title: Effect of Nutritional Counseling Associated With Transcranial Direct-current Stimulation in Binge Eating Reduction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Wolnei Caumo, Professor, surgery departament, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-0206
Record Dates: First submitted 2019-07-02; First posted 2020-01-13 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Transcranial Direct Current Stimulation; Binge-Eating Disorder; Cognitive Behavioral Therapy
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Only the tDCS intervention was masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- a-tDCS and nutritional counseling (Experimental): a-tDCS and nutritional counseling
  Interventions: Combination Product: a-tDCS and nutritional counseling
- s-tDCS and nutritional counseling (Active Comparator): s-tDCS and nutritional counseling
  Interventions: Combination Product: s-tDCS and nutritional counseling
- a-tDCS (Active Comparator): a-tDCS
  Interventions: Device: a-tDCS
- Nutritional counseling (Active Comparator): Nutritional counseling
  Interventions: Behavioral: Nutritional Counseling

INTERVENTIONS:
Device: a-tDCS — Anodal Transcranial direct current stimulation (tDCS) stimulation. Anode will be allocated at DLPFC right and cathode at DLPFC left. The stimulation will occur for 20 min in the intensity of 2 milliampere (mA).
  Arms: a-tDCS
Behavioral: Nutritional Counseling — Presentation delivered through video clip during 20 minutes based on Cognitive Behavioral Therapy interventions
  Arms: Nutritional counseling
Combination Product: a-tDCS and nutritional counseling — a-tDCS + Nutritional Counseling
  Arms: a-tDCS and nutritional counseling
Combination Product: s-tDCS and nutritional counseling — s-tDCS + Nutritional Counseling
  Arms: s-tDCS and nutritional counseling

SUMMARY:
Binge eating disorder is the most prevalent eating disorder, with consequences not only economic but also social. It is related to a set of cognitive alterations related to impulsivity, cognitive function, attention, decision making, emotional control and physiological alterations in the Central nervous system (CNS) in the processing of rewards, mainly in the frontal cortical regions. Psychotherapies are the standard reference treatments, with Cognitive Behavioral Therapy (CBT) being the most indicated nonpharmacological intervention. However, the avoidance rates and the rates of non responders to treatment are significant. In view of this, it is believed that therapeutic approaches aimed at the modulation of the CNS, such as Transcranial direct-current stimulation (tDCS) may have a beneficial effect on the neurobiology of the processes that govern these disorders, thus adding to the effects of CBT and amplifying the therapeutic response.

ELIGIBILITY:
Inclusion Criteria:

* literate
* right - handed individuals
* body mass index ≥ 25 kg / m2
* meet the criteria of the Statistical Diagnostic Manual of Mental Disorders 5th edition (DSM - V) for Binge eating (4 to 7 episodes of binge eating per week).

Exclusion Criteria:

* Pregnancy
* shift workers
* treatment for weight loss in the last 30 days
* bariatric surgery
* formal contraindication for tDCS

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Binge Eating Scale (BES) | 20 minutes
  The Binge Eating Scale is a sixteen item questionnaire used to assess the presence of binge eating behavior indicative of an eating disorder. The questions are based upon both behavioral characteristics (e.g., amount of food consumed) and the emotional, cognitive response, guilt or shame. Each question has 3-4 separate responses assigned a numerical value. The score range is from 0-46= Non-binging (less than 17); Moderate binging (18-26); Severe binging (27 and greater).
Short latency intracortical inhibition | 40 minutes
  Cortical excitability reflects a balance between inhibitory and facilitatory neuronal circuits projected through pyramidal tract output tracts. Transcranial magnetic simulation (TMS) applied to the primary motor cortex (M1) has become widely utilized to assess cortical physiology using paired-pulse paradigms. Preceding subthreshold conditioning stimulus (CS) inhibits the excitability of the motor cortex, which is named short-interval intracortical inhibition (SICI). SICI is a standard method to estimate excitability in a GABAA-ergic circuit in the human cortex;

SECONDARY OUTCOMES:
% Weight loss change | 5 minutes
  % Weight loss change over the treatment
% Reduction of waist circumference | 5 minutes
  % Reduction of waist circumference over the treatment
Three Factor Eating-Questionnaire (TFEQ-R21) | 15 minutes
  TFE-Q access three dimensions of human eating behavior:
  Uncontrolled eating (UE) = Assesses the tendency to lose control over eating when feeling hungry or when exposed to external stimuli. Number of items (NI): 9. Lowest and highest possible raw scores(LH): 9-36.
  Cognitive Restraint (CR) = Assesses the tendency to control food intake in order to influence body weight and body shape. NI: 6. LH: 6-24.
  Emotional Eating (EE)= Measure the propensity to overeat in relation to negative mood states. NI: 6. LH: 6-24.
  We will use the TFEQ-21. The average obtained from the sum of the questions for each domain was converted to a scale ranging from 0 to 100. Higher scores indicate more uncontrolled, restraint and emotional eating.
State and Trait Food Craving Questionnaire (FCQ) | 40 minutes
  The FCQ-T consists of 39 statements and was developed to access food cravings aspects over time and in various situations, considering them as a (usual) trait behavior of the respondent. Higher scores in this questionnaire are related to a more exaggerated eating. Higher scores in this questionnaire are related to a more exaggerated eating.
  The FCQ-S is composed of 15 statements and is a tool sensitive to changes in contextual, psychological and physiological states in response to specific situations (such as stressful events or food deprivation), considering the food craving as a (sporadic) state behavior of the respondent. Higher scores in this questionnaire are associated with greater food deprivation, negative eating-related experiences and a greater susceptibility to triggers that lead to eating.
  Totals of both tools for the full subscales and their dimensions are calculated by adding the corresponding scores of each statement.
Intracortical Facilitation | 40 minutes
  Transcranial magnetic stimulation (TMS) is a magnetic stimulation that can induces in the brain (or in spinal roots, or in nerves) electric currents that can depolarize neurons or their axons. The measures of this technic allow a comprehensive evaluation of the functional state of the corticospinal pathway useful for investigating both physiologic and pathologic conditions. TMS can be used to evaluate excitatory/inhibitory intracortical circuits and to provide information on brain physiology and pathophysiology of various neuropsychiatric diseases as well as on the mechanisms of brain plasticity Intracortical facilitation (ICF) is one of the facilitatory neurophysiological measures of the TMS and is thought to be mainly associated with glutamate receptor-mediated excitatory functions in the motor cortex. We don't have and data with Binge Eating Disorder and is extremely important as it is an indirect measure of Glutamate.
Go/No-go | 20 minutes
  measures impulse control by the ability to inhibit instigated, "prepotent" responses. The task manipulates response prepotency by presenting a preliminary go or no-go cue before the actual go or no-go target is displayed. The cues provide information concerning the probability that a go or no-go target will be presented. The cue-target relationship is manipulated so that the cues have a high probability of correctly signaling a go or no-go target (valid cues), and a low probability of incorrectly signaling a target (invalid cues). Valid cues tend to facilitate response inhibition and speed response execution, whereas invalid cue cues tend to impair response inhibition and slow response execution.
Leptin | 5 minutes
  Leptin is a hormone predominantly made by adipose cells and the small intestine that helps to regulate energy balance by inhibiting hunger. It is an measure of homeostatic eating and considered an obesity biomarker.
Silent period | 40 minutes
  Intracortical inhibition can also be assessed by measurement of the cortical silent period (CSP), which is the interruption of electromyography (EMG) activity following a suprathreshold TMS pulse. The duration of the CSP is a measure of intracortical inhibition due to activation of GABAB interneurons that synapse on pyramidal neurons. We don't have and data with Binge Eating Disorder and is extremely important as it is an indirect measure of gamma-aminobutyrate (GABA).

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, PHD, Study Director — UFRGS and Hospital de Clínicas de Porto Alegre (HCPA)
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Kessler RM, Hutson PH, Herman BK, Potenza MN. The neurobiological basis of binge-eating disorder. Neurosci Biobehav Rev. 2016 Apr;63:223-38. doi: 10.1016/j.neubiorev.2016.01.013. Epub 2016 Feb 2. PMID 26850211
- [Background] Imperatori C, Fabbricatore M, Farina B, Innamorati M, Quintiliani MI, Lamis DA, Contardi A, Della Marca G, Speranza AM. Alterations of EEG functional connectivity in resting state obese and overweight patients with binge eating disorder: A preliminary report. Neurosci Lett. 2015 Oct 21;607:120-124. doi: 10.1016/j.neulet.2015.09.026. Epub 2015 Sep 26. PMID 26409786
- [Background] Peat CM, Berkman ND, Lohr KN, Brownley KA, Bann CM, Cullen K, Quattlebaum MJ, Bulik CM. Comparative Effectiveness of Treatments for Binge-Eating Disorder: Systematic Review and Network Meta-Analysis. Eur Eat Disord Rev. 2017 Sep;25(5):317-328. doi: 10.1002/erv.2517. Epub 2017 May 3. PMID 28467032
- [Background] Fluckiger C, Meyer A, Wampold BE, Gassmann D, Messerli-Burgy N, Munsch S. Predicting premature termination within a randomized controlled trial for binge-eating patients. Behav Ther. 2011 Dec;42(4):716-25. doi: 10.1016/j.beth.2011.03.008. Epub 2011 May 27. PMID 22035999
- [Background] Val-Laillet D, Aarts E, Weber B, Ferrari M, Quaresima V, Stoeckel LE, Alonso-Alonso M, Audette M, Malbert CH, Stice E. Neuroimaging and neuromodulation approaches to study eating behavior and prevent and treat eating disorders and obesity. Neuroimage Clin. 2015 Mar 24;8:1-31. doi: 10.1016/j.nicl.2015.03.016. eCollection 2015. PMID 26110109
- [Derived] Elkfury JL, Antunes LC, Weydmann G, Menegassi LN, Medeiros LF, Cardinal TM, Tocchetto BF, Torres ILS, Fregni F, Bizarro L, Caumo W. The effect of transcranial direct current stimulation and nutritional counseling therapy on attentional bias to food cues: A randomized clinical trial. Clin Nutr ESPEN. 2025 Dec 26;72:102886. doi: 10.1016/j.clnesp.2025.102886. Online ahead of print. PMID 41456817